CLINICAL TRIAL: NCT03134352
Title: A Multi-center, Randomized, Double-blind, Parallel, Placebo Controlled Phase II Study to Evaluate the Efficacy and Safety of Fugan Ointment (ZL-3101) in Subjects With Subacute Eczema
Brief Title: Study to Evaluate the Efficacy and Safety of ZL-3101 in Subjects With Subacute Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zai Lab Pty. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZL-3101-001
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Eczema
Keywords: subacute
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZL-3101(Fugan) bid group (Experimental): Fugan AM + Fugan PM
  Interventions: Drug: ZL-3101
- ZL-3101(Fugan) qd group (Experimental): Fugan AM + Placebo PM
  Interventions: Drug: ZL-3101; Drug: Placebo
- placebo group (Placebo Comparator): Placebo AM + Placebo PM
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZL-3101 — A brown ointment, 10g/tube, 0.4g herb/g ointment, Topical
  Other Names: Fugan ointment
  Arms: ZL-3101(Fugan) bid group; ZL-3101(Fugan) qd group
Drug: Placebo — A brown ointment, 10g/tube, 0.02 g herb/g ointment (5% of Fugan active ointment), Topical
  Arms: ZL-3101(Fugan) qd group; placebo group

SUMMARY:
This is a double-blind, randomized, placebo-controlled multi-center phase IIA study to evaluate the clinical efficacy and safety of Fugan ointment versus placebo applied to involved skin of subjects with mild to moderate subacute eczema.

DETAILED DESCRIPTION:
In this study, patients will be recruited and randomized in a ratio of 2:2:1 into Fugan bid group (Fugan AM + Fugan PM), Fugan qd group (Fugan AM + Placebo PM), and placebo group (Placebo AM + Placebo PM). Randomization will be stratified by disease severity (mild IGA=2 vs. moderate IGA=3).

The patients will be given 3-week treatment and followed up for two weeks after the treatment.

Screening period is set as 1 week. Subjects will be given 3-week treatment and followed up for two weeks after the treatment.

Approximately 310 subjects will be randomized to achieve 250 evaluable subjects completing the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 65 years of age inclusive, at the time of signing the informed consent; from outpatient clinic;
2. Subjects with a diagnosis of subacute eczema (Zhao 2001). Subacute eczema is often developed from improperly treated acute eczema or a few with presented subacute eczema from early on-set. Subacute eczema usually presents with papule, excoriations, crusting and pruritus. Occasionally patient will present with papulovesicle, blister and erosion. Patients also need to meet the requirement of:

   * Subjects must have body surface area (BSA) disease involvement between 3-10% (inclusive) as assessed by palm method;
   * IGA score of 2 or 3;
   * Skin lesions should be on the trunk or extremities, without palms/soles, face/scalp, and vulvar areas involved;
3. Based on TCM theory (Zheng 2002), patients with TCM "damp - heat" symptoms to be included. It is subject to TCM investigator's assessment, and symptoms could be (but not limited to):

   * Main symptoms: erythema, pruritus, papule with less exudation;
   * Secondary symptoms: Mild infiltration, excoriations, crusting, papulovesicle, blister, irritability, thirst, yellowish urine and dry stool;
   * Tongue and pulse analysis: red tongue with yellow or yellowish coating, slippery pulse model;
4. Subjects are general in good health; except for eczema, there are no other health conditions that possibly interfere with the study results;
5. A signed and dated written informed consent is obtained from the subject.

Exclusion Criteria:

1. The subject presents with or has the history of any systemic disorders or active skin diseases (e.g. psoriasis) that would in any way confound interpretation of the study results;
2. The subject has a current complication of overt bacterial, fungal or viral infection for which treatment with anti-infective are indicated;
3. Have the history of hepatic and kidney function insufficiency, hepatic dysfunction ALT or AST>1.5 ULN, kidney function BUN, Cr>1.5 ULN;
4. QT interval corrected according to Bazett's formula or QT interval corrected according to Fridericia's formula ≥450 msec; or QTc ≥480 msec in subjects with bundle branch block;
5. Have the history or examination verified by physical and screening of clinically significant cardiovascular, pulmonary, gastrointestinal, liver, renal, hematological, neurological, abnormalities and psychology disorders which will interfere with the efficacy and/or safety of the individual subject;
6. History of allergy to any component of test medications to be used in the study;
7. The subject has been exposed to below therapy within the set timeframe:

   * Systemic administration of anti-histamine agents 1 week
   * Systemic administration of corticosteroid 4 weeks;
   * Topical corticosteroid agents administered in the diseased skin 1 week;
   * Systemic administration of immunosuppressive drugs 4 weeks;
   * Topical immunosuppressive drugs administered in the diseased skin 1 week;
   * Systemic administration of any TCM drugs 2 weeks;
   * Topical administration of any TCM drugs 1 week;
   * UV therapy 4 weeks

   The use of inhaled/intranasal steroids is permitted prior to and during the conduct of the study if already being used by the subject.
8. The subject has a past history of alcohol or drug abuse;
9. Pregnant women (as confirmed by a positive urine human chorionic gonadotrophin (HCG) test), women who are breast feeding, or sexually active women of child bearing potential who are not practicing an acceptable method of birth control (birth control pill, patch, implant, barrier with spermicidal jelly, IUD, etc.), as determined by the investigator. An acceptable method of birth control must be used during the entire study in sexually active women of childbearing potential. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant. Abstinence is considered as a medically acceptable form of contraception;
10. The subject has received an investigational drug or participated in any other research trial within 30 days;
11. Other subjects that investigator deemed as unsuitable for the trial;
12. Subject's EASI score reaches 2 and above for lichenification and/or edema.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) score changes from baseline to day 21 | 21 days
  To evaluate efficacy of Fugan ointment applied to involved skin of subjects with mild to moderate subacute eczema

CONTACTS AND LOCATIONS:
Overall Officials: Bin Li, Principal Investigator — Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of TCM
Locations (6):
- China (6):
  - Beijing Hospital of Traditional Chinese Medicine, Beijing
  - Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing
  - Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing
  - Jiangsu Province Hospital of Traditional Chinese Medicine, Nanjing
  - Shanghai Dermatology Hospital, Shanghai
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of TCM, Shanghai

IPD SHARING:
Plan to Share IPD: No